CLINICAL TRIAL: NCT02565862
Title: A Drug-drug Interaction Study Between the Novel Anti-hepatitis c Virus (HCV) Agent Daclatasvir and The Antidiabetic Agent Metformin in Healthy Volunteers
Brief Title: A Drug-drug Interaction Study Between Daclatasvir and Metformin
Acronym: DATE-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 14.11
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis C; Diabetes Mellitus; Insulin Resistance
Keywords: HCV; Diabetes Mellitus; Daclatasvir; Metformin; drug-drug interaction; pharmacokinetics
MeSH Terms: conditions — Hepatitis C; Diabetes Mellitus; Insulin Resistance | interventions — daclatasvir; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Active Comparator): Day 1-2: 500mg twice daily (BID) metformin film-coated tablets
  Day 3-8: 1000mg BID metformin film-coated tablets
  Interventions: Drug: Metformin
- Treatment B (Experimental): Day 15-16: 500mg BID metformin film-coated tablets + 60mg once daily (QD) daclatasvir film-coated tablets
  Day 17-22: 1000mg BID metformin film-coated tablets
  + 60mg QD daclatasvir film-coated tablets
  Interventions: Drug: Daclatasvir; Drug: Metformin

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: Daklinza
  Arms: Treatment B
Drug: Metformin

SUMMARY:
This study aims to provide clinical information on a potential drug-drug interaction between daclatasvir and metformin.

DETAILED DESCRIPTION:
Daclatasvir is a recently approved anti-HCV agent that is a cytochrome P450 3a (CYP3A) substrate but does not affect CYP3A itself. It is also a moderate inhibitor of various membrane transporters such as organic anion-transporting polypeptide 1B1 (OATP1B1) , p-glycoprotein (P-gP), and organic cation transporter (OCT) 1 and 2.

Metformin is used to treat diabetes mellitus. It is an OCT-2 and OCT-1 substrate and when combined with daclatasvir increased levels of metformin may occur, with risk on hypoglycaemic episodes. The Summary of Product Characteristics (SmPC) of daclatasvir currently does not mention this potential drug-drug interaction.

HCV is associated with insulin resistance (IR) which may develop to diabetes mellitus (DM). The prevalence of IR in HCV infected patients is estimated varying from 30% to 70%. Several studies showed that IR has a negative impact on the achievement of an undetectable HCV viral load after completing 12 weeks of treatment (Sustained Virologic Response (SVR)).

This study aims to provide clinical information on a potential drug-drug interaction between daclatasvir and metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 and not older than 55 years at screening.
2. Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to Day 1.
3. Subject has a Quetelet Index (Body Mass Index) of 18 to 35 kg/m2, extremes included.
4. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, and electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
6. Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

1. Creatinine clearance below 60mililiter/minute (ml/min).
2. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
3. Positive HIV test.
4. Positive hepatitis B or C test.
5. Pregnant female (as confirmed by an Human chorionic gonadotropin (hCG) test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
6. Therapy with any drug (for two weeks preceding Day 1), except for acetaminophen (max 2 gram/day).
7. Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders (increased alanine aminotransferase (ALAT)/ASAT), hormonal disorders (especially diabetes mellitus), coagulation disorders.
8. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
9. History of or current abuse of drugs, alcohol or solvents.
10. Inability to understand the nature and extent of the study and the procedures required.
11. Participation in a drug study within 60 days prior to Day 1.
12. Donation of blood within 60 days prior to Day 1.
13. Febrile illness within 3 days before Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | up to 24 hours after administration for daclatasvir and up to 12 hours after administration for metformin

SECONDARY OUTCOMES:
adverse events | 4 weeks
  adverse events will be collected up to 4 weeks in total (entire study)

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- CRCN, Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Smolders EJ, Colbers A, de Kanter CTMM, Velthoven-Graafland K, Wolberink LT, van Ewijk-Beneken Kolmer N, Drenth JPH, Aarnoutse RE, Tack CJ, Burger DM. Metformin and daclatasvir: absence of a pharmacokinetic-pharmacodynamic drug interaction in healthy volunteers. Br J Clin Pharmacol. 2017 Oct;83(10):2225-2234. doi: 10.1111/bcp.13323. Epub 2017 Jun 6. PMID 28474741